CLINICAL TRIAL: NCT01991119
Title: Efficacy of Propafenone Versus Dronedarone for the Maintenance of Sinus Rhythm in Patients With Atrial Fibrillation After DC Cardioversion
Brief Title: Efficacy of Propafenone Versus Dronedarone for the Maintenance of Sinus Rhythm in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Keun On, Principle investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-03-085-001
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Propafenone; Dronedarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone; Dronedarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propafenone (Active Comparator): Propafenone group
  Interventions: Drug: Propafenone
- Dronedarone (Active Comparator): Dronedarone group
  Interventions: Drug: Dronedarone

INTERVENTIONS:
Drug: Propafenone
  Arms: Propafenone
Drug: Dronedarone
  Arms: Dronedarone

SUMMARY:
the purpose of this study is to compare the ability of propafenone and dronedarone to maintain sinus rhythm after DC cardioversion

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmia requiring continuous therapy. Conversion to and maintenance of sinus rhythm is important. Propafenone and dronedarone has been used as treatment for maintenance of sinus rhythm after DC cardioversion. But there are no direct comparison study.

The purpose of this study is to compare the ability of propafenone and dronedarone to maintain sinus rhythm after DC cardioversion.

ELIGIBILITY:
Inclusion Criteria:

* a patient with persistent atrial fibrillation who received successful DC cardioversion

Exclusion Criteria:

* prior amiodarone use
* NYHA class III or IV heart failure
* Left ventricular ejection fraction < 35%
* second or third AV block
* sick sinus syndrome
* heart rate < 50 beat per minute
* myocardiac infarction within 3 months
* pregnant women
* severe hepatic dysfunction
* QT prolongation > 500ms or PR interval > 180ms
* history of hypersensitivity for drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Young Keun On, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Cardiac and Vascular Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Chun KJ, Byeon K, Im SI, Park KM, Park SJ, Kim JS, On YK. Efficacy of dronedarone versus propafenone in the maintenance of sinus rhythm in patients with atrial fibrillation after electrical cardioversion. Clin Ther. 2014 Sep 1;36(9):1169-75. doi: 10.1016/j.clinthera.2014.07.013. Epub 2014 Aug 16. PMID 25134972